CLINICAL TRIAL: NCT04687514
Title: Effects of Glucagon-Like Peptide-1 Analogs on Sexuality - a Randomized, Double-blind, Placebo-controlled Trial With Crossover Design
Brief Title: Effects of Glucagon-Like Peptide-1 Analogs on Sexuality
Acronym: DESIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Goldschmidt-Jacobson Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2020-02572; me20ChristCrain3
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Sexual Functioning
Keywords: dulaglutide; Glucagon-like peptide-1 (GLP-1) analogs; Massachusetts General Hospital - Sexual Functioning Questionnaire (MGH-SFQ); GLP-1 receptor
MeSH Terms: interventions — dulaglutide

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled trial with crossover design: Dulaglutide or placebo weekly subcutaneously for 4 weeks; in random order, separated by washout period of at minimum 28 days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, health-care providers and data collectors are blinded to treatment allocation. Excluded from the blinding are defined study nurses administrating the injections as injection devices (dulaglutide/ placebo) are not identical. The unblinded study nurses are otherwise not involved in the trial. During the injection participants are blindfolded such as the injection device and the injection site is not visible for them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase a (V1a-Ev2a): Dulaglutide first- Phase b (V1b-Ev2b) Placebo second (Experimental): Dulaglutide is injected via pen s.c. once a week. The titration scale will be 1x 1.5mg in 0.5 ml in the first week and 2x 1.5 mg in 2x 0.5 ml once weekly for 3 further weeks. Dulaglutide or placebo weekly subcutaneously for 4 weeks; in random order, separated by washout period of at minimum 28 days.
  Interventions: Drug: Dulaglutide; Drug: Placebo
- Phase a (V1a-Ev2a): Placebo first- Phase b (V1b-Ev2b) Dulaglutide second (Experimental): The Placebo will be injected via syringe and contains 0.5ml (only first injection) or 2x0.5ml (second to fourth injection) of 0.9% sodium chloride (0.9% NaCl). Dulaglutide or placebo weekly subcutaneously for 4 weeks; in random order, separated by washout period of at minimum 28 days.
  Interventions: Drug: Dulaglutide; Drug: Placebo

INTERVENTIONS:
Drug: Dulaglutide — Dulaglutide: first week 1x 1.5mg in 0.5 ml, following 3 weeks 2 x 1.5 mg weekly in 0.5ml each, via Pen s.c.
Drug: Placebo — Placebo: first week 1x0.5 ml physiological saline (0.9% sodium chloride) injection s.c. via syringe, following weeks 2x0.5 ml physiological saline (0.9% sodium chloride) injection s.c. via syringe once weekly for 3 further weeks.

SUMMARY:
This placebo-controlled, double-blind crossover study is to evaluate the GLP-1 analogue dulaglutide regarding changes in sexuality, the mood and the reproductive axis in healthy men.

DETAILED DESCRIPTION:
This placebo-controlled, double-blind crossover study is to evaluate the GLP-1 analogue dulaglutide regarding changes in sexuality, the mood and the reproductive axis in healthy men.

The study consists of following two phases:

* Phase a (V1a-Ev2a): baseline evaluation (V1a), application of the trial medication (dulaglutide or placebo) during 4 weeks (V1a-V4a), evaluation of the primary and secondary outcomes (V2a-V4a, Ev1a), followed by a washout period of at minimum 28 days before evaluation of the last secondary outcome (Ev2a) and cross-over
* Phase b (V1b-Ev2b): baseline evaluation (V1b), application of the trial medication (dulaglutide or placebo) during further 4 weeks (V1b-V4b), evaluation of the primary and secondary outcomes (V2b-V4b, Ev1b), followed by a washout period of at minimum 28 days before evaluation of the last secondary outcome (Ev2b) and study end after study termination visit (STV).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men with normal weight (BMI 18.5-25kg/m2 or BMI 25.1-30kg/m2 and waist circumference <102cm)
* Written informed consent
* Active sex life (sex with partner or masturbation ≥2x/week)
* Satisfactory sex life
* No Hypogonadism (morning total testosterone ≥12mmol/l)

Exclusion Criteria:

* History of pancreatitis
* History of psychiatric disease (by questioning the participant, also regarding current psychiatric treatment)
* Daily nicotine abuse
* Alcohol consumption (>1 glass/day)
* Substance abuse (as eg cannabis, anabolic steroids, benzodiazepines, opiates, psychostimulants)
* Regular intake of medication at any time

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Change in sexual functioning, assessed with the German version of the Massachusetts General Hospital - Sexual Functioning Questionnaire (MGH-SFQ). | at baseline (before start of treatment) and after each week of treatment (V1, V2, V3, V4 and EV1), up to 10 weeks.
  Change in sexual functioning, assessed with the German version of the Massachusetts General Hospital - Sexual Functioning Questionnaire (MGH-SFQ). The MGH-SFQ consists of five items addressing libido, arousal, orgasm, erection, overall sexual satisfaction. Each item is rated by a discrete score ranging from 1 to 6 (1 = greater than normal; 2 = normal; 3 = minimally diminished; 4 = moderately diminished; 5 = markedly diminished; 6 = totally absent). The MGH-SFQ sum score ranges from 5 to 30, with 10 indicating normal functioning, values < 10 indicating improved functioning, and values > 10 indicating diminished functioning. The primary endpoint is the absolute change from baseline to end of treatment in the MGH-SFQ sum score. A positive score change indicates worsening of sexual functioning. The primary endpoint will be compared for a difference between verum and placebo.

SECONDARY OUTCOMES:
Mood changes, assessed by the German Version of the Patient Health Questionnaire-9 for Depression (PHQ-9) | at baseline and after end of treatment (V1 and EV1), up to 10 weeks.
  Mood changes, assessed by the German Version of the Patient Health Questionnaire-9 for Depression (PHQ-9). . Each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day).
Change in hormones of the reproductive axis | at baseline and after end of treatment (V1 and EV1), up to 10 weeks.
  Change in hormones of the reproductive axis (total testosterone (measured), free testosterone (derived from total testosterone), luteinizing hormone (LH), follicle stimulating hormone (FSH), sex hormone binding globulin (SHBG), prolactin and oxytocin.)
Change in semen concentration | at baseline and eight weeks after end of treatment
  Change in semen concentration
Change in semen motility | at baseline and eight weeks after end of treatment
  Change in semen motility

OTHER OUTCOMES:
Change in weight (kg) | at baseline and after end of treatment (V1 and EV1), up to 10 weeks.
  Change in weight (kg)
Change in BMI | at baseline and after end of treatment (V1 and EV1), up to 10 weeks.
  Change in BMI
Change in HbA1c | at baseline and after end of treatment (V1 and EV1), up to 10 weeks.
  Change in HbA1c
Change in serum glucose | at baseline and after end of treatment (V1 and EV1), up to 10 weeks.
  Change in serum glucose
Change in adverse event (AE)-survey | at Visit 2, Visit 3, Visit 4 and Evaluation Visit (up to 4 weeks)
  Change in AE-survey (following symptoms will be assessed: abdominal pain, nausea, vomitus, diarrhoea, local irritation or pain, allergic reaction, fatigue, light-headedness)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Winzeler, Dr. med., Principal Investigator — Endocrinology, Diabetes and Metabolism, University Hospital Basel
Locations (1):
- University Hospital Basel, Endocrinology, Diabetes and Metabolism, Basel, Switzerland